CLINICAL TRIAL: NCT00255684
Title: Non-Myeloablative Conditioning and Unrelated Umbilical Cord Blood Transplantation for Children and Adults With Serious Oncohematologic Diseases
Brief Title: Fludarabine, Cyclophosphamide, and Total-Body Irradiation Followed by Cyclosporine and Mycophenolate Mofetil in Treating Patients Who Are Undergoing a Donor Umbilical Cord Blood Transplant for Hematologic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000448637; URCC-U19403; URCC-RSRB-10063
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: graft versus host disease; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; acute undifferentiated leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia; chronic myelomonocytic leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; juvenile myelomonocytic leukemia; primary myelofibrosis; refractory hairy cell leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; refractory chronic lymphocytic leukemia; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); de novo myelodysplastic syndromes; recurrent mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent mantle cell lymphoma; relapsing chronic myelogenous leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; recurrent adult Hodgkin lymphoma; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Juvenile; Primary Myelofibrosis; Leukemia, Hairy Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Recurrence; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous; Dendritic Cell Sarcoma, Interdigitating | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conditioning therapy followed by TBI (Experimental): Fludarabine, Cyclophosphamide; Total-Body Irradiation Followed by Cyclosporine and Mycophenolate Mofetil
  Interventions: Biological: graft-versus-tumor induction therapy; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: umbilical cord blood transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: graft-versus-tumor induction therapy
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: umbilical cord blood transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and cyclophosphamide, and radiation therapy before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation followed by cyclosporine and mycophenolate mofetil works in treating patients who are undergoing a donor umbilical cord blood transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency, extent, and rate of donor (myeloid and lymphoid) engraftment in patients with serious hematologic malignancies treated with nonmyeloablative conditioning regimen comprising fludarabine, cyclophosphamide, and low-dose total-body irradiation followed by unrelated allogeneic umbilical cord blood transplantation and post-transplant immunosuppression comprising cyclosporine and mycophenolate mofetil.
* Correlate clinical and umbilical cord blood-related factors with engraftment in patients treated with this regimen.
* Determine transplant-related complications, in terms of toxicity, myelosuppression, infections, and acute and chronic graft-versus-host disease, in patients treated with this regimen.
* Determine disease-free and overall survival of patients treated with this regimen.
* Determine treatment-related mortality of patients treated with this regimen.

OUTLINE: This is a uncontrolled, pilot study.

* Nonmyeloablative conditioning regimen: Patients receive fludarabine IV over 30 minutes daily on days -6 to -2 and cyclophosphamide IV over 2 hours on day -6 and undergo low-dose total-body irradiation (TBI) on day 0.
* Unrelated allogeneic umbilical cord blood transplantation (UCBT): After completion of TBI, patients undergo 1 or 2 unrelated allogeneic UCBTs on day 0.
* Post-transplant immunosuppression: Patients receive oral or IV cyclosporine daily beginning on day -3 and continuing until day 180 and oral or IV mycophenolate mofetil twice daily on days 0-30.

Patients are followed periodically for 1 year after transplantation.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia (AML) with or without history of myelodysplastic syndromes, meeting 1 of the following criteria:

    * In first complete remission (CR-1) with unfavorable cytogenetics and/or achieved CR-1 after ≥ 1 course of induction therapy
    * Secondary or treatment-related AML
    * In second or further complete remission
    * Relapsed with ≤ 20% blasts in the bone marrow AND no circulating blasts
  * Acute lymphoblastic leukemia (ALL), meeting 1 of the following criteria:

    * In CR-1 with unfavorable cytogenetics or elevated WBC at presentation OR failed to achieve CR-1 after ≥ 4 weeks of induction therapy
    * In second or further complete remission
    * Relapsed with ≤ 20% blasts in the bone marrow AND no circulating blasts
  * Other acute leukemic variants allowed at the discretion of the principal investigator
  * Chronic myelogenous leukemia (CML), meeting 1 of the following criteria:

    * In first chronic phase AND refractory to or unable to tolerate imatinib mesylate
    * In second or further chronic phase
    * In first or second accelerated phase
  * Myelodysplastic syndromes with intermediate 2- or high-risk International Prognosis Scoring System (IPSS) score, including any of the following:

    * Refractory anemia
    * Refractory anemia with excess blasts
    * Chronic myelomonocytic leukemia
  * Myeloproliferative disorders with poor prognosis, including any of the following:

    * Myelofibrosis with myeloid metaplasia

      * No ≥ grade 3 myelofibrosis
    * Atypical CML
    * Juvenile myelomonocytic leukemia
  * Other clonal hemopathies with an accepted poor prognosis
  * Multiple myeloma with chromosome 13 abnormalities and/or progression after prior autologous bone marrow transplantation (BMT)
  * Chronic lymphocytic leukemia, meeting 1 of the following criteria:

    * Primary refractory OR relapsed and refractory disease (less than partial remission)
    * Relapsed twice on or after prior chemotherapy
  * Lymphoma, meeting both of the following criteria:

    * Hodgkin's or non-Hodgkin's lymphoma in > CR-1 OR failed primary induction
    * Chemosensitive disease, defined as > 50% reduction in mass size after the most recent chemotherapy
* Must meet ≥ 1 of the following criteria:

  * Over 45 years of age
  * Has undergone prior autologous or allogeneic BMT
  * Charlson^ comorbidity score ≥ 2
* Must have a high degree of tumor control (salvage therapy allowed)
* At high risk for treatment-related mortality with a myeloablative conditioning regimen
* No massive splenomegaly

  * Patients may become eligible after splenectomy or radiotherapy to the spleen
* No 5/6 or 6/6 HLA-matched related donor available
* No well-matched (i.e., ≥ 9/10 HLA match by high-resolution typing) unrelated donor available

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Transaminases ≤ 4 times ULN (unless due to underlying disease)

Renal

* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* Ejection fraction ≥ 30%

Pulmonary

* DCLO ≥ 35%

Other

* Negative pregnancy test
* No uncontrolled viral, bacterial, or fungal infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Other

* At least 3 months since prior immunosuppressive therapy
* At least 10 days since prior salvage therapy for patients not in at least morphologic or radiologic complete remission

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-12; Primary Completion 2013-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon L. Phillips, MD, Principal Investigator — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Conditioning Therapy Followed by TBI: Fludarabine, Cyclophosphamide; Total-Body Irradiation Followed by Cyclosporine and Mycophenolate Mofetil
  graft-versus-tumor prophylaxis therapy
  cyclophosphamide
  cyclosporine
  fludarabine phosphate
  mycophenolate mofetil
  umbilical cord blood transplantation
  radiation therapy
Period: Overall Study
Arm/Group | Conditioning Therapy Followed by TBI
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Conditioning Therapy Followed by TBI
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived 100 Days or Longer
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Conditioning Therapy Followed by TBI
Number analyzed (Participants) | 16
participants | 13

2. Secondary Outcome: Number of Participants Who Developed Acute Graft Versus Host Disease
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Conditioning Therapy Followed by TBI
Number analyzed (Participants) | 16
participants | 0

ADVERSE EVENTS:
Arm/Group | Conditioning Therapy Followed by TBI
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Therapy Followed by TBI (N=16)
graft versus host disease (Immune system disorders) | 3
multi-organ failure (General disorders) | 2
Post-transplant lymphoproliferative disorder (Immune system disorders) | 1
Syndrome of Inappropriate Antidiuretic Hormone Secretion (Metabolism and nutrition disorders) | 1
sepsis (Infections and infestations) | 3
relapsed transplant resulting in death (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes